CLINICAL TRIAL: NCT04924387
Title: Effects of a Procedure Programme in Patients With Non-specific Low Back Pain. Comparative Intervention Based on Therapeutic Exercise, Therapeutic Exercise With Kinesio Tape and Manual Therapy Prior to the Therapeutic Exercise
Brief Title: Manual Therapy and Exercise in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2019-2020/138
Record Dates: First submitted 2020-10-19; First posted 2021-06-14 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
Keywords: chronic pain; manipulation, musculoskeletal; catastrophisation; kinesiotaping; exercise
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Motor Activity | interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The groups will be arranged randomly and the masking technique to be used will the double blind procedure. The subjects will be randomly selected through the GPower 3.1 programme. The random allocation to each group will be made just by one external researcher, this way, neither the main researcher, nor the participants, will know their allocation. Furthermore, the inspector who will collect the evaluation data won't know either the allocation of each subject.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (EXP group) (Experimental): The experimental group (EXP Group) is going to follow a programme of stabilisation through specific therapeutic exercises of the lumbopelvic centre. Two weekly sessions will be programmed for 12 weeks, making a total of 24 sessions. Each sesión will have a duration of 60 minutes, the first 5 minutes for a warm-up and the last 10 for a cool-down phase of active stretching. All patients will start learning how to activate the abdominal muscles in the first training session. The exercise progression will be adapted according to the capacity of each patient, considering their pain levels. The exercices will be made in 1 to 3 series of among 8 and 15 repetitions and the isometric contractions for 5 to 10 seconds. The rests between series will be of 30 seconds, and between exercies of 2-3 minutes.
  Interventions: Procedure: Exercise
- Experimental Group and Manual Therapy (MT Group) (Active Comparator): Additionally to the core exercises previously exposed in Group EXP, Group MT will lay on the stretcher first, where the physiotherapist will work on a manual therapy thrust. The patient will receive an impulse technique in lateral decubitus position, with high velocity and low range on both sides.
  Interventions: Procedure: Exercise
- Experimental Group and Kinesio Tape (KT Group) (Active Comparator): The experimental group plus kinesio tape (KT Group) will go previously through physiotherapy, where a kinesio tape band will be applied (kinesio tape "Nondolens" 5cm x 5cm black color), in Y technique, by applying the KT base in neutral position of the lumbar spine without any tension on the tape.
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — All patients will start learning how to activate the abdominal muscles in the first training session. The exercise progression will be adapted according to the capacity of each patient, considering their pain levels. The exercises will be made in 1 to 3 series of among 8 and 15 repetitions and the isometric contractions for 5 to 10 seconds. The rests between series will be of 30 seconds, and between exercises of 2-3 minutes.
  Other Names: musculoskeletal manipulation; kinesiotaping

SUMMARY:
Non-specific low back pain is one of the main causes of disability for health care worldwide. The effectiveness of therapeutic exercise, of kinesio tape and of manual therapy in the treatment of low back pain is evaluated, but not a comparison of these techniques. Moreover, can these techniques be combined?

DETAILED DESCRIPTION:
Non-specific low back pain is one of the main causes of disability for health care worldwide. Nowadays, the mostly used technique to research low back muscular activity is electromyography.

Among the published studies, the effectiveness of therapeutic exercise, of kinesio tape and of manual therapy in the treatment of low back pain is evaluated, but not a comparison of these techniques.

The main objective that is aimed by this thesis, is the evaluation of muscular activation in the reduction of non-specific low back pain through a 12 weeks procedure programme, which includes therapeutic exercise combined with other treatment techniques, and assessing the psycho-social characteristics of pain.

This study's population will be composed by at least 16 individuals per group, both male and female, with ages among 20 and 80.

Participants will be randomly and blindly divided in three groups of intervention. The three groups will be: the experimental group or EXP Group (all participants subject to therapeutic exercise), the experimental group, which will also be subject to manual therapy (MT Group) and finally, the experimental group, which will also be subject to kinesio tape work (KT Group).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with low back pain.
* Patients who are in Stage 1 of the Oswestry scale.
* Not receiving pharmacological treatment such as anti-inflammatories or corticosteroids
* Be able to understand the exercises and spanish language.

Exclusion Criteria:

* Having any back surgery.
* Be taking any medication at the time of the study.
* Have a pathology in which exercise is contraindicated (spondylolisthesis, spondylolysis, spondyloarthrosis).
* Be in a state of gestation or if there is the possibility of being.
* Present or have presented some oncological process.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Oswestry | (12 weeks)
  The Oswestry (ODI) test will be made to all participants at three months. The results of this scale will provide the necessary information to know the degree of symptomatology of the patient and will therefore help in the planification and procedure to the patient. That is why, it has been established that all participants in Stage 1 of the test are subsidiaries to make all the treatment modes of the study (manual therapy and exercise). This way, we are able to rise the homogeneity that imposes a diagnostic label such as the chronic low back pain.

SECONDARY OUTCOMES:
Kinesiophobia (TKS) | (12 weeks)
  The mostly used questionnaire to evaluate kinesiophobia is the TKS (Tampa Kinesiophobia Scale) questionnaire, which we will use to measure which is the fear to movement of patients of low back pain. This scale includes work related lesions, lesions due to repetitive effort, relapses and the avoidance-fear. The questionnaire is composed of 17 items in which there is a differentiation between the negative an positive elements.
  This questionnaire will be filled in based on a Likert scale which ranges between 0 and 5, being 0 never and 5 always. The total punctuation ranges between 17 and 68, the higher the rate, the higher the degree of kinesiophobia.
Catastrophism (PCS) | (12 weeks)
  To quantify the degree of catastrophism in the present study, the validated spanish version will be used as the pain catastrophism scale (PCS). The PCS is a 13-item self-report scale of 13 items, that presents same factor structure composed of the factors of rumination, despair and magnification. For each of these factors, it is given a value of 0 (without agreement) to 4 (always), so that at the end the examiner obtains a score between 0 and 52. Low scores indicate a low level of catastrophism and high values show high levels of catastrophism.
Self-efficacy: questionnaire | (12 weeks)
  To assess self-efficacy, it will be used the Chronic Pain Self-Efficacy Questionnaire, which assesses a person's belief in their ability to perform a specific behavior. It consists of 19 items, a Likert-type scale and a response range of 0 to 10, where 0 is equivalent to feeling totally incapable, 5 moderately incapable and 10 fully capable. The result determines that the higher the score, the greater the degree of self-efficacy.
Visual analog scale (VAS) | (12 weeks)
  The VAS from 0 to 100, the scale considered to be the most representative, with the VAS being the best option due to its easy understanding and handling. This scale constitutes an effective tool to subjectively quantify this range, more discriminating than the scale that establishes its values from 0 to 10. This way, 0 will be considered as non-existent pain reflected by the individual and 10 as the worst pain imaginable by the patient.
Pressure algometry | (12 weeks)
  Pressure algometry is considered a useful method to calculate the degree of sensitization of deep tissues. It will be carried out using an algometer, which in this study will consist of a manometer attached to a cylindrical rubber tip. The manometer measures the pressure applied through the rubber and the patient should signal when this pressure starts being painful. This way, it will be established the pressure pain threshold (PPT). Algometry is a widely studied and validated technique to quantify sensitivity in the diagnosis of symptomatic points and myofascial trigger points. The reliability of pressure algometry is relatively high, presenting coefficients of 0.9 and 0.95.
Electromyography | (12 weeks)
  to obtain an objective measure of the muscle activation, surface electromyography will be used to evaluate the main core muscles - basically the transverse abdomen.
  The electromyograph to be used will be the FREEEMG model of the brand BTS Bioengineering. It is a wireless electromyograph with probes attached to the prefilled electrodes, which collect the information. No additional hardware is required, as the same software processes the information taken. The data resolution is 16 bit and the acquisition frequency of 1 kHz.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Vicente Mampel, Phd, Study Director — Fundación Universidad Católica de Valencia San Vicente Mártir
Locations (1):
- FundacionUCV, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992